CLINICAL TRIAL: NCT06369220
Title: A Study of the Clinical Utility of Point of Care Cobas® Liat CT/NG/MG Nucleic Acid Test Versus Current Standard Practice
Brief Title: A Study of the Cobas® Liat CT/NG/MG Test Versus Current Standard Practice for Managing Participants at Increased Risk of Sexually Transmitted Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Molecular Systems, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LIA-STI-542
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chlamydia Trachomatis Infection; Neisseria Gonorrhoeae Infection; Mycoplasma Genitalium Infection
Keywords: Sexually transmitted infections; Urogenital infections; Point of care testing
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard of Care (SOC) Arm: Standard Practice (Other): In the SOC arm, the clinician will evaluate the participant based on standard practice.
  Interventions: Other: Standard of Care (SOC): Clinician's Standard Practice
- Point of Care (POC) Arm: cobas® liat CT/NG/MG (Experimental): In the POC arm, the clinician will evaluate the participant and will be provided POC test results upon which they may choose to base their clinical decisions.
  Interventions: Diagnostic Test: cobas® liat CT/NG/MG nucleic acid test

INTERVENTIONS:
Diagnostic Test: cobas® liat CT/NG/MG nucleic acid test — The cobas® CT/NG/MG nucleic acid test for use on the cobas® Liat® System is an investigational, automated, qualitative in vitro nucleic acid diagnostic test that utilizes real-time polymerase chain reaction (PCR) for the direct detection of Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Mycoplasma genitalium (MG) nucleic acid in male/female urine and vaginal swabs (clinician-collected and self-collected) in cobas® PCR Media.
  Arms: Point of Care (POC) Arm: cobas® liat CT/NG/MG
Other: Standard of Care (SOC): Clinician's Standard Practice — Standard of care (SOC) is defined as the traditional/typical diagnosis and treatment steps in practice recommended by the CDC guidelines that rely upon clinical syndromic presentations and/or external laboratory testing.
  Arms: Standard of Care (SOC) Arm: Standard Practice

SUMMARY:
This study is designed to assess the comparative clinical utility of the point of care cobas® liat CT/NG/MG to current standard practices in the diagnosis and treatment of urogenital infections with Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Mycoplasma genitalium (MG).

DETAILED DESCRIPTION:
The study is designed as a block randomized, controlled 2-arm prospective study. The study targets to enroll approximatively 348 participants at increased risk of sexually transmitted infections (STIs)-participants who have known contact with CT/NG/MG (including participants who report knowledge or suspicion of STI exposure, despite the uncertainty of the specific STI pathogen or contact testing results), or participants with symptoms suggestive of STI-to participate in this study. Participants who give consent will provide demographic information and urogenital specimen(s) for CT/NG/MG testing on the cobas® liat system and for external laboratory-polymerase chain reaction (EL-PCR) testing. Participants will be randomized in a 1:1 ratio in blocks (of multiples of 2) stratified by the site to either of the following arms:

* Standard of Care (SOC)
* Point of Care (POC)

In both arms, the clinician will see and evaluate the participant and will complete a standardized form, known as a patient management plan (PMP), at the conclusion of the participant's encounter. The critical difference between the arms is that the clinician in the POC arm will be provided POC test results upon which they may choose to base their clinical decisions, whereas the SOC arm will not receive POC test results.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active people
* People seeking medical services for symptoms consistent with a sexually transmitted infection (STI) and/or known exposure to an STI

Exclusion Criteria:

* Previously enrolled in the study
* Unable to provide informed consent
* Currently pregnant
* Declines POC testing
* Presents for routine STI screening (asymptomatic)
* Use of antimicrobial agents active against CT, NG, or MG during the 21 days before sample collection. Example of such antimicrobial agents include the following: Macrolides (e.g., azithromycin and erythromycin); Penicillins (e.g., amoxicillin); Tetracyclines (e.g., doxycycline); Fluoroquinolones (e.g., ciprofloxacin, ofloxacin, levofloxacin, and moxifloxacin); Cephalosporins (e.g., ceftriaxone and cefixime)
* Use of phenazopyridine-containing urinary pain relief medicines (ie, Azo or Pyridium) within 2 days prior to sample collection
* Use of any over-the-counter feminine hygiene products (internally or externally), such as vaginal moisturizers, lubricants (e.g., Replens, RepHresh, etc.), and feminine washes/vaginal douches, etc. within the 3 days prior to sample collection. The use of tampons or pads during menses is not an exclusionary criterion.
* Contraindication to vaginal swab sampling where vaginal swab sampling is the only option available
* Urination within 1 hour prior to sample collection (for subjects providing urine sample)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Given Inappropriate Treatments for All Pathogens Combined (CT, NG, and MG) | On the day of the medical encounter (Day 1)
  An inappropriate treatment is defined as under and/or overtreatment on the day of the medical encounter based on CDC recommendations for the pathogen-specific results obtained by EL-PCR.

SECONDARY OUTCOMES:
Percentage of Participants Given Inappropriate Treatment for CT Infection | On the day of the medical encounter (Day 1)
Percentage of Participants Given Inappropriate Treatment for NG Infection | On the day of the medical encounter (Day 1)
Percentage of Participants Given Inappropriate Treatment for MG Infection | On the day of the medical encounter (Day 1)
Mean Satisfaction and Confidence Rating Scores of SOC and POC, According to Healthcare Professionals' Responses to the CSDT Questionnaire | Once every 2 weeks until end of study (approximately 4 months)
  Healthcare professionals will rate their confidence in and their satisfaction with the POC test and SOC procedures on a 5-point scale from very confident to very unconfident and on a 5-point scale from very satisfied to very dissatisfied, respectively, in response to the Clinician Satisfaction with Diagnostic Test Questionnaire (CSDT-Q).
Mean Satisfaction Rating Scores of SOC and POC, According to Participants' Responses to the PSDT Questionnaire | On the day of the medical encounter (Day 1)
  Participants will rate their satisfaction with the POC test and SOC procedures on a 5-point scale from very satisfied to very dissatisfied in response to the Patient Satisfaction with Diagnostic Test Questionnaire (PSDT-Q).

CONTACTS AND LOCATIONS:
Overall Officials: Zune Huynh, MD, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - San Francisco City Clinic, San Francisco, California
  - Planned Parenthood of Northern, Central, and Southern New Jersey, Inc., Hamilton Square, New Jersey
  - Planned Parenthood of Northern, Central and Southern New Jersey, Perth Amboy, New Jersey
  - Baylor Scott & White Health - Kileen, Killeen, Texas

IPD SHARING:
Plan to Share IPD: No